CLINICAL TRIAL: NCT04698564
Title: Utility of Hyperpolarized 13C-pyruvate Metabolic Magnetic Resonance Imaging in the Diagnosis and Risk-Stratification of Prostate Cancer
Brief Title: Utility of Hyperpolarized 13C-pyruvate Metabolic Magnetic Resonance Imaging
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18149GCCC ; HP-00084316
Record Dates: First submitted 2020-10-01; First posted 2021-01-07 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single-arm study in patients who are suspected or known to have prostate cancer (Experimental): Perform metabolic magnetic resonance imaging on men suspected to have a prostate cancer to understand if metabolic MRI can be safely performed on this population
  Interventions: Drug: Hyperpolarized 13C-Pyruvate

INTERVENTIONS:
Drug: Hyperpolarized 13C-Pyruvate — Hyperpolarized Pyruvate (13C) Injection, containing spin-polarized ("hyperpolarized") [ 13C]pyruvate, is being studied as a diagnostic agent in combination with 13C spectroscopic MR imaging. The aim is to visualize [13C]pyruvate and its metabolites and thereby distinguish between anatomical areas with normal vs. abnormal metabolism, which should be useful in diagnosing and characterizing, for example, malignancy.
  Hyperpolarized Pyruvate (13C) Injection and [13C]pyruvate are general terms used throughout this brochure, that refer to all 13C labeling patterns, such as [1- 13C]pyruvate, [2- 13C]pyruvate and [1,2- 13C]pyruvate. From biological and safety standpoints, pyruvate with each of the labeling patterns behaves identically in the human body [Koletzko et al., 1997].

SUMMARY:
This is a two-tiered pilot study in which there will be no randomization and no placebo treatment. This study will be to perform metabolic magnetic resonance imaging on men suspected to have a prostate cancer to understand if metabolic MRI can be safely performed on this population

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than 40 and less than 80 years
2. Clinical suspicion or history of prostate cancer reflected by one of the following:

   * PSA > 4ng/ml
   * Abnormal DRE exam
   * Known tissue diagnosis of prostate cancer from prior workup
3. Patient planning to undergo either a MRI targeted biopsy or radical prostatectomy for prostate cancer workup or treatment

Exclusion Criteria:

1. Inability to undergo MRI scan
2. Inability to receive IV contrast as per institutional protocol.

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
CTCAE v4.0 higher than grade 2 | Within three years post treatment
  Quantify the number of participants who get this scan and have treatment-related adverse events as assessed by CTCAE v4.0 higher than grade 2. Determine the number of participants who successfully complete a scan which meets a minimum quality standard as measured by signal to noise ratio on the scan.
  hyperpolarized metabolic MRI in the diagnosis of prostate cancer.

SECONDARY OUTCOMES:
Accuracy of metabolic MRI to diagnose prostate cancer | Within three years post treatment
  To study the accuracy of hyperpolarized metabolic MRI to diagnose prostate cancer. Compare the prediction of cancer from the MRI scan compared to actual diagnosis of cancer by any subsequent workup or procedure the participant undergoes. Prediction of cancer from MRI scan will be performed by assigning a standardized score (PIRADS v2.0). Actual diagnosis of cancer will be based on tissue pathology (with cancer grade characterized using the prostate cancer ISUP Grade Group system) from any procedure the patient undergoes.
Utility of metabolic MRI over standard MRI imaging in the diagnosis of prostate cancer | Within three years post treatment
  To examine the added utility of metabolic MRI over standard MRI imaging. Quantify the number of participants in which the MRI provided extra information that otherwise was not available during the course of the patient's workup.
Correlative metabolic analysis of tissue metabolite concentrations versus cancer diagnosis | Within three years post treatment
  To perform correlative metabolic analysis related to cancer diagnosis. Using the research tissue when it is available. Analyze tumor samples when available from participants and characterize the metabolite concentration (microgram/mg of tissue) within the tumor to determine how the concentration value compares to two outcomes of interest: 1: the numerical suspicion score (PIRADS v2.0 system) from the imaging from the patient and 2: The presence of cancer and grade of cancer (ISUP Grade Group system), when present, from pathology analysis performed on the tissue from the patient available. Analyze tumor samples when available from participants and characterize the metabolite concentration within the tumor to determine how this compares to the information from the imaging from the patient and pathology analysis performed on the tissue

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland Medical Center, Baltimore, Maryland, United States